CLINICAL TRIAL: NCT05496647
Title: The Effect Of Vırtual Realıty, Musıc Therapy, And Stress Ball Applıcatıon On Paın And Anxıety Durıng Daıly Gynecologıcal Surgery
Brief Title: Vırtual Reality, Music Therapy and Stress Ball-related Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Nurdan Demirci, PhD RN, Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MarmaraU-OZ-2022
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Pain; Anxiety
Keywords: Nursing; Virtual Reality; Music Therapy,; Stress Ball; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Masking Description: Criteria for Inclusion in the Research
  * Over 18 years old,
  * Can speak Turkish,
  * Subjected to daily gynecological surgery for the first time,
  * Does not have any psychiatric disease and mental perception problems,
  * Having no vision, hearing, and perception problems,
  * Having no physical problems squeezing a stress ball,
  * There will be women who agree to participate in the research verbally and in writing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Reality (VR) (Experimental): Virtual Reality Application (VR) VR group patients will be shown VR videos that include landscapes such as nature and the sea, giving people a feeling of comfort and peace, and making them feel like they are inside. During the surgical procedure, VR videos will be watched for an average of 20 minutes with X-brand VR glasses. In the research, similar studies will be examined and 360o VR video, which is a licensed product with atmospheric music background, containing relaxing nature images and nature sounds will be used.
  Interventions: Other: Virtual Reality
- Music Therapy (Experimental): Music Therapy Application During the surgical procedure, an mp3 player, and music therapy CDs of uşşak and Hüseyni will be used. (Oline will also create a list from music platforms (fizzy-Spotify, etc.)) Before starting the procedure, the patients will be asked about their music preferences and the music will be played to the patients (20 minutes) during the procedure in line with their preferences. Headphones provided by the researcher will be used for patients with headphones, and for patients without headphones.
  The music authorities used (hüseyni and uşşak) will be provided and used by order, by obtaining the necessary permissions from the official site of TÜMATA.
  Interventions: Other: Music Therapy
- Stress Ball Application (Experimental): Stress Ball Application A sufficient number of stress balls will be provided by the investigator for each patient to use separately before starting the study. Before starting the day-to-day gynecological surgery, patients in the stress ball group will be given a round, colored, medium-hard, compressible Knaftmed ball made of high-quality silicone. To avoid implying that the procedure is inherently stressful, it will be referred to as a squeezing ball when instructing patients about stress ball application.
  During the surgical procedure, it will be said that he can squeeze the stress ball as often as he wants for about 20-25 minutes and the stress ball will be given to each patient.
  Interventions: Other: Stress Ball Application
- Control (Experimental): During the process; Women in the control group will not undergo any intervention other than routine surgery.
  Interventions: Other: Control

INTERVENTIONS:
Other: Virtual Reality — Before the surgical procedure; the Structured Patient Description Form, Fear of Pain Scale, Life Information Follow-up Form, State Anxiety Inventory, and Visual Comparison Scale forms will be filled by the researcher using a face-to-face interview technique with the woman.
  During the process; the Preferred video will be watched with Virtual Reality Glasses for approximately 20 minutes during the process, After Daily Gynecological Surgery 1. Measurements; Immediately after the procedure, within the first 10 minutes; Life Information Follow-up Form, Visual Comparison Scale will be filled.
  2. Measurements After Daily Gynecological Surgery; At the 1st hour after the procedure, Vital Information Follow-up Form and Visual Comparison Scale will be filled.
  3. Measurements After Daily Gynecological Surgery; In the 2nd hour after the procedure; Life Information Follow-up Form, State Anxiety Inventory, Visual Comparison Scale and Satisfaction Evaluation Form will be filled.
  Arms: Virtual Reality (VR)
Other: Music Therapy — Before the surgical procedure; the Structured Patient Description Form, Fear of Pain Scale, Life Information Follow-up Form, State Anxiety Inventory, and Visual Comparison Scale forms will be filled by the researcher using a face-to-face interview technique with the woman.
  During the process; During the procedure, the preferred music for Music Therapy will be played for approximately 20 minutes, After Daily Gynecological Surgery 1. Measurements; Immediately after the procedure, within the first 10 minutes; Life Information Follow-up Form and Visual Comparison Scale will be filled.
  2. Measurements After Daily Gynecological Surgery; In the 1st hour after the procedure, the Vital Information Follow-up Form and Visual Comparison Scale will be filled.
  3. Measurements After Daily Gynecological Surgery; In the 2nd hour after the procedure; Life Information Follow-up Form, State Anxiety Inventory, Visual Comparison Scale, and Satisfaction Evaluation Form will be filled.
  Arms: Music Therapy
Other: Stress Ball Application — Before the surgical procedure; the Structured Patient Description Form, Fear of Pain Scale, Life Information Follow-up Form, State Anxiety Inventory, and Visual Comparison Scale forms will be filled by the researcher using a face-to-face interview technique with the woman.
  During the process; the Stress ball will be played for approximately 20 minutes during the process.
  After Daily Gynecological Surgery 1. Measurements; Immediately after the procedure, within the first 10 minutes; Life Information Follow-up Form and Visual Comparison Scale will be filled.
  2. Measurements After Daily Gynecological Surgery; In the 1st hour after the procedure, the Vital Information Follow-up Form and Visual Comparison Scale will be filled.
  3. Measurements After Daily Gynecological Surgery; In the 2nd hour after the procedure; Life Information Follow-up Form, State Anxiety Inventory, Visual Comparison Scale, and Satisfaction Evaluation Form will be filled.
  Arms: Stress Ball Application
Other: Control — Before the surgical procedure; the Structured Patient Description Form, Fear of Pain Scale, Life Information Follow-up Form, State Anxiety Inventory, and Visual Comparison Scale forms will be filled by the researcher using a face-to-face interview technique with the woman.
  During the process; Women in the control group will not undergo any intervention other than routine surgery.
  After Daily Gynecological Surgery 1. Measurements; Immediately after the procedure, within the first 10 minutes; Life Information Follow-up Form and Visual Comparison Scale will be filled.
  2. Measurements After Daily Gynecological Surgery; In the 1st hour after the procedure, the Vital Information Follow-up Form and Visual Comparison Scale will be filled.
  3. Measurements After Daily Gynecological Surgery; In the 2nd hour after the procedure, the Life Information Follow-up Form, State Anxiety Inventory, Visual Comparison Scale, and Satisfaction Evaluation Form will be filled.
  Arms: Control

SUMMARY:
Outpatient surgical interventions; It is defined as surgical applications where the application time is short, the risk of complications is low, there is no need for intensive care after the intervention, and the patients can be discharged on the same day. It is applied in areas such as otolaryngology and maxillofacial surgery. Among all these areas, gynecological surgery is the area where the most outpatient surgery is performed. Some of the gynecological procedures that are generally applied in day surgery are as follows; Colposcopy, hysteroscopy, laparoscopy, dilatation-curettage, laparoscopic tubal ligation, treatment of the cervix with cautery or laser, removal of vulvar cysts, laser conization, cervical polypectomy and removal of Bartholin cysts.

In many state hospitals in our country, in daily gynecological surgical procedures; in some cases by premedication, in some cases under local anesthesia; however, patients are usually processed without anesthesia.

Virtual Reality, which is a type of computer system using human-machine interfaces, has been used in pain and anxiety management in different applications in many areas known as painful medical procedures in recent years.

Music therapy is defined as "the systematic use of music in a therapeutic relationship aimed at improving, maintaining and advancing emotional, physical and mental health". Music therapy has important physiological effects that reduce heart rate, blood pressure, body temperature, and respiratory rate, distract attention, increase the quality of life of patients, and reduce pain.

Stress ball emerges as a simple, reliable, inexpensive, and easily accessible method that helps patients reduce their anxiety. Squeezing the stress ball during the surgical procedure allows patients to have direct control over the object, increasing feelings of empowerment. In this way, it has a positive effect on anxiety and patient satisfaction without interfering with the surgical procedure. Based on all these reasons; The aim of this study is to determine the effects of virtual reality, music therapy, and stress ball applications on vital signs, pain, anxiety, and patient satisfaction during daily gynecological surgery.

DETAILED DESCRIPTION:
Virtual Reality

Virtual Reality (VR) is a term formed from the words virtual and reality. According to the Turkish Language Association; Virtuality, which means unreal, or hypothetical, derives from the Latin word "virtual". The reality is; the real is defined as the whole of the things that exist and the truth. Virtual reality, which emerged as a concept in the 1950s, started to be used in application areas in the 1900s.

Virtual reality, which has been used only for space and military research as a computer-based, high-cost technology for years, has recently become widespread in the fields of medicine, education, entertainment, librarianship, museology, architecture, and industrial design with different applications developed for mobile devices.

Today, common and easily accessible android-based smart devices capable of running virtual reality are used. The image is obtained using a combination of framed simple optical lenses that hold the phone at a fixed distance perpendicular to the user's gaze direction. The working system of three-dimensional resuscitation devices is based on stereographic vision properties. After the relevant applications are installed on the smartphone, the device divides the screen into two, and thanks to the acquisition of different images for the right and left eyes, the illusion of the spatial existence of three-dimensional animated objects is obtained.

Virtual Reality is a simulation model that gives a sense of reality to its participants, is created based on computers, and allows mutual communication.

Virtual Reality Application in Pain and Anxiety Management

Virtual reality, which is a type of computer system using human-machine interfaces, has been used in the management of pain and anxiety in many different applications known as painful medical procedures in recent years. According to the researchers' hypotheses, virtual reality; acts as a non-pharmacological method using cognitive and attentional processes on the body's complex pain modulation system. Although its neurobiological mechanisms have not been fully explained, studies have interestingly reported that it brings positive results in pain management.

In virtual reality applications, patients feel that they are in the image, their attention is effectively distracted from the pain, and the perception of pain is reduced. In recent years, virtual reality as a distraction application; It is used in the management of pain and anxiety in procedures such as burn debridement, injection applications, wound care, toothache, endoscopy procedure, phantom, and chronic pain, and chemotherapy applications.

Music Therapy in Pain and Anxiety Management

Music therapy is a method that has been used frequently among complementary and alternative medicine applications for centuries. Music, which consists of regular, harmonious rhythms and sounds that we hear with our ears, is a behavior that expresses the aesthetics found in human nature. The therapeutic use of music has an active role in making people feel and communicate with their emotional dimension.

The first scientific theorist of the use of music therapy in treatment was Pythagoras. Today, a quintuple scale system is known as the 'Pythagorean Scale' or the 'Fiddler Scale'. For the ancient Greeks, music is considered the most basic element of spiritual education and purification of the soul from evil. Athennoaops aimed to alleviate the pain by playing an instrument in the area of pain by using the vibration effect. In Turkish-Islamic Civilization; According to great philosophers and scientists such as İbn-i Sina and Farabi, music not only improves the hearing power, but also the cognitive ability of people with the suggestions it creates. Music was also used in the treatment of mental illnesses with the melodies made by the Sufis who were dealing with Sufi music. XV-XVI. between the Kayseri Gevher Nesibe Medical Madrasa and Edirne Sultan II. The architecture of Ottoman-era hospitals such as the Bayezid Hospital was built in accordance with the isolation of patients, ventilation, and treatment with music.

Today, the effectiveness of music therapy as a complementary medicine application has been proven in many studies. American Music Therapy Association; reported that music significantly reduced pain and anxiety levels. There are studies stating that music is effective in pain during burn dressing and cancer-related pain, reduces opioid use after surgery, reduces the stress levels of patients during childbirth and different medical applications, and decreases blood pressure and pulse values.

music therapy; By focusing the patients on the rhythm of the music, distracts their attention from the pain, and activating the door control system, reduces the perception of pain. Music therapy increases the secretion of endorphins and relaxes the individual. music therapy; is used in the treatment of pain and anxiety as a non-pharmacological method that is easy to apply, economical, and has no side effects.

Stress Ball in Pain and Anxiety Management

A stress ball is a simple, reliable, inexpensive, and easily accessible method that helps reduce the anxiety of patients. It is stated that the use of stress balls generally relieves patients.

A stress ball, which is one of the distraction methods, is also an effective method in providing cognitive focus. It is seen in studies that stress ball application is used to reduce the anxiety and pain of patients. Squeezing a stress ball during the surgical procedure allows patients to have direct control over the object in their palm and increases patients' feelings of empowerment. Applying a stress ball in this way has a positive effect on anxiety and patient satisfaction without interfering with the surgical procedure. In another study; It has been found that holding a stress ball reduces both pain and anxiety in patients undergoing surgical procedures.

In the study of Yanes et al. to evaluate the effects of a stress ball or hand holding on pain, anxiety, and satisfaction in skin cancer surgery performed under local anesthesia, it was concluded that anxiety decreased in all groups. In the study, it was concluded that the stress ball helped reduce anxiety in patients who were anxious before the procedure. In the study conducted by Kasar et al. on hemodialysis patients, it was concluded that the use of a stress ball has a positive effect on stress.

In the study conducted to determine the effect of distraction methods used during the cystoscopy procedure on pain, anxiety, and satisfaction, it was concluded that the level of post-procedural anxiety was lower in the intervention groups (music, video, and stress ball) than the control group, and the satisfaction was higher.

In a randomized controlled study in which three different non-pharmacological methods (coughing technique, spirometer blowing, and stress ball squeezing) were evaluated in reducing pain during intravenous catheterization; It was concluded that the pain averages of the patients in the coughing technique, spirometer blowing and stress ball groups were lower than the control group.

In another study examining the effectiveness of distraction methods for pain and anxiety management during invasive venous surgery, it was concluded that pain and anxiety were significantly lower in the interaction with nurses and the stress ball group.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Can speak Turkish,
* Subjected to daily gynecological surgery for the first time,
* Does not have any psychiatric disease and mental perception problems,
* Having no vision, hearing, and perception problems,
* Having no physical problems squeezing a stress ball,
* There will be women who agree to participate in the research verbally and in writing.

Exclusion Criteria:

* Having used analgesic or anesthetic drugs within 24 hours before or during the procedure
* Using antidepressant, anxiolytic and sedative drugs
* Communication difficulties and mental disability
* Patients with severe vision and hearing problems, and physical disabilities (with open wounds on their hands, insufficient muscle strength to squeeze a stress ball) will not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who will undergo daily gynecological surgery
Enrollment: 160 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 5 Months
  Fear of Pain Scale-III; Participants mark the option that best describes the severity of their fear according to their pain experiences regarding the items listed on the scale. In the scoring, it means that 1- fear is never heard, and 5-fear is excessive. The lowest score that can be obtained in total is 30, and the highest score is 150.The lowest score that can be obtained for the sub-dimensions is 10, and the highest score is 50. The higher the individual's score on the scale, the higher the fear of pain.
  Visual Analog Scale = VAS; In order to determine the severity of the pain experienced by the participants during and after the outpatient gynecological surgical procedure, score measurements in centimeters (cm) will be determined on the vertically prepared GCS. Visual Comparison Scale (0cm;No pain, 0.5cm- 3.0cm;Mild pain, 3.5cm-6.5cm;Moderate pain, 7.0cm-10.0cm;Severe pain).

SECONDARY OUTCOMES:
Anxiety Intensity | 5 Months
  The State Anxiety Inventory (STAI-S) will be used to measure the instantaneous anxiety levels before and after the surgical procedure, and the anxiety levels of the individuals will be determined. According to the results obtained, while the average anxiety scores are between 36 and 41, above this value indicates high anxiety level and below this value indicates low anxiety level.
Patient Information Form | 5 Months
  Identifiable Information used by the sender is one of the first methods to be implemented. This section consists of education-training-gynecological 30th section such as age, educational status, educational status, social education.
Life Information Tracking Form | 5 Months
  In the measurement of vital signs of individuals, devices that measure digital blood pressure and pulse, O2 saturation will be used by applying the necessary hygiene rules at patient transitions.
Patient Satisfaction Evaluation Form | 5 Months
  Form, prepared by the researchers in line with the literature, consists of 11 questions questioning the satisfaction status of Virtual Reality, Music Therapy and Stress Ball applications, and a chart that starts with dissatisfaction (0) and shows the level of satisfaction (10).

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba öz, PhD RN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)